CLINICAL TRIAL: NCT00456690
Title: Endocrine and Nutritional Assessment in B Thalassemia Major - A Clinical Trial
Brief Title: Endocrine and Nutritional Assessment in B Thalassemia Major
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5190906/2.EMC
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Thalassemia
Keywords: Thalassemia; Nutrition; Endocrine; BMI
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Thalassemia Mayor Patients
  Interventions: Other: Nutritional recommendations

INTERVENTIONS:
Other: Nutritional recommendations — Nutritional status assessment including complete endocrine and lipid laboratory profile and after one year of nutritional follow up a secondary assessment will be done

SUMMARY:
B Thalassemia patients developed short stature and low weight in spite no evident endocrine abnormalities. One hypothesis is that they developed some degree of malnutrition,then the purpose of this study is to assess the nutritional status before nutritional intervention and after one year. Siblings of the patients will serve as a control group.

BMI, lipid and endocrine profile and leptin levels will be analysed in the study group only.

DETAILED DESCRIPTION:
The nutritionist will advice the patients about calories requirement and intake, balance diet and follow up the patients during the study period of one year. No special medicaments or drug therapy will be provided as part of the study protocol

ELIGIBILITY:
Inclusion Criteria:

* All patients above age 5 ys treated in the clinic.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2007-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
BMI | 1 year study

CONTACTS AND LOCATIONS:
Overall Officials: Carina Levin, MD, Principal Investigator — Pediatric Hematology Unit, Ha'Emek Medical Center; Ariel Koren, MD, Study Director — Pediatric Hematology Unit - Ha'Emek Medical Center
Locations (1):
- Pediatric Hematology Unit - HaEmek Medical Center, Afula, Israel